CLINICAL TRIAL: NCT04965948
Title: Evaluation of the Anti-inflammatory Effects of a Snack Enriched With Camelina Sativa Oil in Free-living Older Adults: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effects of Camelina Sativa Oil in Free-living Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14012021; E47F17000020009 (Other: Grantor or Funder: Regione Lombardia - POR FESR 2014-2020)
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Inflammation; Malnutrition; Hyperglycemia; Dyslipidemias
Keywords: Inflammaging; Healthy aging; Older Adults; Omega-3 fatty acid; Camelina Sativa; Inflammation; Micronutrients deficiency
MeSH Terms: conditions — Inflammation; Malnutrition; Hyperglycemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Snack enriched with camelina sativa oil
  Interventions: Other: Novel food snack
- Placebo group (Placebo Comparator): Snack no enriched with camelina sativa oil
  Interventions: Other: Placebo snack

INTERVENTIONS:
Other: Novel food snack — Consumption of snack enriched with camelina sativa oil, twice a day for 12 weeks
  Arms: Active group
Other: Placebo snack — Consumption of placebo snack (no enriched with camelina sativa oil), twice a day for 12 weeks
  Arms: Placebo group

SUMMARY:
The present study aims at evaluating the anti-inflammatory effects of a novel food in older adult volunteers. Briefly, this randomized, double-blind and placebo-controlled study is performed on 91 apparently healthy older adults (age≥65 years) before and after 12 weeks' consumption of a snack enriched with camelina Sativa oil. Subjects were randomized into two groups (active group vs placebo group).

DETAILED DESCRIPTION:
Ninety-one volunteers (26M/65F) are enrolled according to the following inclusion criteria i) free-living older adults ≥ 65 years; ii) apparently healthy subjects; iii) subjects who do not take vitamin supplements/integration and/or omega 3 polyunsaturated fatty acids; iv) subjects without food allergies.

All volunteers are informed about the purpose of the study and the potential risk and provide their informed consent.

Subjects are randomized into two groups: active group (13M/36F) vs placebo group (13M/29F).

The main objective of this project is to test the efficacy of the 12-weeks consumption of a novel food (snack enriched with camelina Sativa oil) on the inflammatory status in older adults.

The primary and secondary endpoints are:

i) Investigation of changes in serum CRP levels and serum levels of pro- and anti-inflammatory cytokines, in the active group (volunteers consumed enriched snack with camelina Sativa oil) and placebo group, after 12 weeks of snacking (T1), compared to baseline (T0) (primary endpoint).

ii) Evaluation of changes in serum lipid panel parameters after the consumption of the novel food in both the active and placebo groups (secondary endpoint).

iii) Evaluation of changes in glucidic status after the consumption of the novel food in both the active and placebo groups (secondary endpoint).

iv) Evaluation of changes in the levels of omega 3 polyunsaturated fatty acids in both the active and placebo groups (secondary endpoint).

v) Evaluation of the nutritional status at T0 and at T1 in both the active and placebo groups (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Age over 65
* Free-living
* No food allergy
* Apparent good health
* Acceptance and sign of informed consent

Exclusion Criteria:

* Age under 65
* Living in a nursing home, extended care
* Hospitalized
* Presence food allergy
* Without acceptance and sign of informed consent
* Taking vitamin supplements/integration and/or omega 3 polyunsaturated fatty acids

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory status evaluation. | Baseline (T0) and after 12 weeks of intervention (T1).
  Investigation of changes in serum CRP levels (pg/mL) and serum levels of pro- and anti- inflammatory cytokines (TNF-α, pg/mL; TGF-beta1, pg/mL and TGF-beta2, pg/mL; IL-18 pg/mL).

SECONDARY OUTCOMES:
Lipid panel parameters evaluation. | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of changes in serum lipid panel parameters (total cholesterol, mg/dL; triglycerides, mg/dL; HDL cholesterol, mg/dL; LDL cholesterol, mg/dL).
Omega 3 polyunsaturated fatty acids evaluation. | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of changes in the levels of omega 3 polyunsaturated fatty acids.
Glucidic profile evaluation -glucose levels | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of changes in the levels of glucose (mg/dL)
Glucidic profile evaluation - insulin levels | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of changes in the levels of insulin (μU/mL).
Glucidic profile evaluation - glycated haemoglobin levels | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of changes in the levels of glycated haemoglobin (mmol/mol).
Glucidic profile evaluation - HOMA index | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of changes in the HOMA index.
Nutritional status evaluation - hepatic function | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of ALT (U/L), AST (U/L).
Nutritional status evaluation - renal function | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of creatinine (mg/dL).
Nutritional status evaluation. | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of prealbumin (g/L).
Nutritional status evaluation - micronutrients | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the calcium (mg/dL), magnesium (mg/dL).
Nutritional status evaluation - micronutrients | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of iron (μg/dL) and zinc (μg/dL)
Nutritional status evaluation - vitamins | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of vitamin B9 (ng/mL) and vitamin D (ng/mL).
Nutritional status evaluation - vitamins | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of vitamin B12 (pg/mL).
Nutritional status evaluation - hyperhomocysteinemia | Baseline (T0) and after 12 weeks of intervention (T1).
  Evaluation of nutritional status by assessing the serum levels of Homocysteine (μM).
Anthropometric parameters evaluation - weight | Baseline (T0).
  Evaluation at baseline of weight (Kg).
Anthropometric parameters evaluation - height and waist circumference | Baseline (T0).
  Evaluation at baseline of height (cm) and waist circumference (cm).
Ponderal status evaluation | Baseline (T0).
  Evaluation at baseline of Body Mass Index (Kg/m2) to investigate the prevalence of overweight or obesity.
Fat distribution evaluation. | Baseline (T0).
  Evaluation at baseline of Waist to height ratio (WHtR) as a proxy of fat distribution and metabolic diseases risk.
Body composition evaluation. | Baseline (T0).
  Evaluation at baseline of reactance (Ohm) and resistance (Ohm) by using vectorial bioimpedance analysis.
Muscle strength evaluation. | Baseline (T0).
  Evaluation at baseline of muscle strength (Kg) by using a handgrip-dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, MD, Prof., Principal Investigator — University of Pavia
Locations (1):
- University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Giuseppe R, Di Napoli I, Tomasinelli CE, Vincenti A, Biino G, Sommella E, Ferron L, Campiglia P, Ferrara F, Casali PM, Cena H. The Effect of Crackers Enriched with Camelina Sativa Oil on Omega-3 Serum Fatty Acid Composition in Older Adults: A Randomized Placebo-Controlled Pilot Trial. J Nutr Health Aging. 2023;27(6):463-471. doi: 10.1007/s12603-023-1925-x. PMID 37357331